CLINICAL TRIAL: NCT00465140
Title: Effects of Creatine Supplementation on Renal Function in Sedentary Healthy Males Urdergoing Aerobic Training: a Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effects of Creatine Supplementation on Renal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EEFEUSP-021284
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: creatine supplementation
Behavioral: aerobic exercise training

SUMMARY:
Creatine (CR) supplementation is commonly used by athletes. However, its effects on renal function remain controversial. The aim of this study was to evaluate the effects of creatine supplementation on renal function and oxidative stress in healthy sedentary males (18-35 years old) submitted to exercise training. Our hipothesis is that creatine supplementation does not affect renal function in this population.

DETAILED DESCRIPTION:
Creatine (CR) supplementation is commonly used by athletes. However, its effects on renal function remain controversial. Purpose: The aim of this study was to evaluate the effects of creatine supplementation on renal function and oxidative stress in healthy sedentary males (18-35 years old) submitted to exercise training. Methods: Subjects (n = 18) were randomly divided in two groups and were allocated to receive treatment with either creatine (CR) (~10g • day-1 over three months) or placebo (PL) (dextrose). All subjects undertook moderate intensity aerobic training, in three 40-minute sessions per week, during 3 months. Serum creatinine, TBARS, serum and urinary sodium and potassium were determined at baseline and at the study endpoint. Furthermore, cystatin C was also assessed prior to training (PRE), after 4 (POST 4) and 12 weeks (POST 12). Results: There were decreased in both oxidative stress (evaluated by TBARS - µM/24 h) (PRE CR: 8.2  4.4; PL: 6.4  0.8 vs. POST 12 CR: 2.5  1.8; PL: 2.1  1.6, p=0.0001) and cystatin C levels (mg/L) (PRE CR:0.82  0.09; PL: 0.88  0.07 vs. POST 12 CR: 0.71  0.06; PL: 0.75  0.09, p=0.0001) over the time, suggesting an increase in glomerular filtration rate. There were no significant differences between groups in other renal parameters investigated. Conclusions: These data indicate that high-dose creatine supplementation throughout three months does not provoke renal dysfunction in sedentary healthy males urdergoing aerobic training. Moreover, our results suggest that moderate aerobic training per se could improve renal function.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary healthy males,
* Euthrofic,
* Age beteween 18-35 y

Exclusion Criteria:

* Food supplement users,
* Pre-existing renal dysfunction,
* Pre-existing cardioavascular disease,
* Subjetcs physically active or athletes,
* Obesity,
* Drugs users

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2004-01; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, ms, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil